CLINICAL TRIAL: NCT01379261
Title: Rapid Endovascular Catheter Core Cooling Combined With Cold Saline as an Adjunct to Percutaneous Coronary Intervention For the Treatment of Acute Myocardial Infarction
Brief Title: Efficacy of Endovascular Catheter Cooling Combined With Cold Saline for the Treatment of Acute Myocardial Infarction
Acronym: CHILL-MI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Philips Healthcare (Industry); Lund University (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHILL-MI
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Myocardial Infarction; Myocardial Reperfusion Injury; Anterior Wall Myocardial Infarction; Inferior Wall Myocardial Infarction
Keywords: STEMI; primary PCI; Hypothermia; Endovascular cooling; Cardiac MRI
MeSH Terms: conditions — Myocardial Infarction; Myocardial Reperfusion Injury; Anterior Wall Myocardial Infarction; Inferior Wall Myocardial Infarction; ST Elevation Myocardial Infarction; Hypothermia | interventions — Cool-Down Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia treatment (Active Comparator): 1-2 liters of cold saline and central venous catheter cooling with Philips InnerCool RTx Endovascular System prior to PCI
  Interventions: Procedure: Cooling
- Standard treatment (No Intervention): Standard treatment

INTERVENTIONS:
Procedure: Cooling — 1-2 liters of cold saline and central venous catheter cooling with Philips InnerCool RTx Endovascular System prior to PCI
  Other Names: Hypothermia
  Arms: Hypothermia treatment

SUMMARY:
The purpose of this study is to determine whether treatment of patients suffering from ST-elevation myocardial infarction (STEMI) with 1-2 liters of cold saline and central venous catheter cooling with Philips InnerCool RTx Endovascular System prior to percutaneous coronary intervention (PCI) result in a reduction in infarct size.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is the leading cause of mortality in the western world today. Although reperfusion of the ischemic myocardium is a prerequisite for myocardial salvage, it has been described that the reperfusion in itself may cause additional damage to the myocardium (reperfusion injury). In the safety & feasibility trial RAPID MI-ICE we demonstrated that treatment of patients suffering from STEMI with 1-2 liters of cold saline and central venous catheter cooling with Philips InnerCool RTx Endovascular System prior to PCI was feasible, safe and resulted in a 38% reduction in infarct size/myocardium at risk. The aim of the present study is to confirm this finding in a larger multicenter trial.

The study is a randomized, controlled, evaluator blinded, multicenter trial enrolling 120 patients at ten sites.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms and signs of myocardial infarction and have a 12-lead ECG providing evidence of an ongoing acute myocardial infarction, involving a large area of myocardium, as defined by the following ECG criteria. The ECG changes should be present upon arrival to the cath lab:

   1. Anterior infarct: ST-segment elevation >0.2mV measured 0.08 sec after the J point in 2 or more anatomically contiguous precordial leads, V1 through V4; and/or >0.2mV in lead V5 V6.
   2. Inferior infarct: ST elevation >0.2mV measured 0.08 sec after the J point in 2 or more anatomically contiguous inferior leads, coupled with ST depression in 2 contiguous anterior leads for a total ST deviation (inferior ST elevation plus anterior ST depression) of >0.8mV.
2. Present to the study PCI lab within six (6) hours of the onset of acute cardiac ischemic signs or symptoms (such as chest pain or pressure, arm or jaw pain, dyspnea, nausea/vomiting, or syncope).
3. Be a candidate for PCI and have PCI planned as the immediate intervention.
4. Be willing and able to comply with study procedures, including returning for the MRI scan at 4 ±2 days and be available for additional follow up Subject understands study procedures and agrees to participate in the study by giving written informed consent.
5. Be in Killips Class I.

Exclusion Criteria:

1. Age less than eighteen (<18) years of age
2. Age greater than or equal to eighty (80) years of age
3. Are pregnant.
4. Having an aortic dissection
5. History of a prior large myocardial infarct or an infarct in the same segment that is currently affected.
6. Acute administration of a thrombolytic agent for the qualifying MI
7. Clinical suspicion of a non-thrombotic (e.g., pericarditis, vasospasm, takotsubo, illicit drug use) cause for ST-segment elevation as determined by the investigator
8. If (during the screening process) the determination is made by site-study personnel that initiation of cooling prior to diagnostic coronary angiography is technically not feasible for any reason (should the patient be randomized to the Hypothermia Arm), the prospective subject should not be enrolled.
9. Known risk for heparin induced thrombocytopenia (HIT)
10. Require an immediate surgical or procedural intervention other than PCI (e.g. CABG)
11. Present in cardiogenic shock or with end-stage cardiomyopathy
12. Have undergone at least ten (10) minutes of cardiopulmonary resuscitation (CPR) prior to presentation to the PCI facility
13. History of surgical coronary artery revascularization (e.g. CABG)
14. Active bleeding, coagulopathy, or other contraindication to the placement of a heparin-coated 14F central venous catheter via a 14F femoral venous introducer sheath (e.g., known history of heparin induced thrombocytopenia, or IVC filter)
15. Contraindications to hypothermia
16. Personal or familial history of malignant hyperthermia
17. Known end-stage renal disease (ESRD; e.g., on dialysis, or status-post renal transplant), known severe hepatic failure (e.g., cirrhosis, or acute hepatitis), or any other contraindication to receiving meperidine (such as use of MAO inhibitors within previous 14 days, history of seizures, history of hypersensitivity to meperidine, etc.).
18. Serious concurrant medical condition likely to result in death during the next 12 months. Any other acute or chronic condition which the Investigator believes will unacceptably increase the risk of study participation or interfere with study procedures and assessments.
19. Contraindication to MRI (e.g., cardiac pacemaker, ICD, nerve stimulator, brain aneurysm clips, cochlear implants, claustrophobia)
20. Deemed unsuitable by the investigators to participate in the study.
21. Active or recent (within 1 month prior to study enrollment) participation in another investigational clinical research study.
22. Enrollment in or planned to be enrolled in another study of AMI therapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size (as a percentage of myocardium at risk) assessed by cardiac MRI. | At 4±2 days

SECONDARY OUTCOMES:
Myocardial infarct size (as a percentage of myocardium at risk) both assessed by cardiac MRI at 4±2 days in the patients who are cooled and achieve a target temperature of < 35 C prior to PCI. | At 4±2 days
Myocardial infarct size (as a percentage of myocardium at risk) both assessed by cardiac MRI at 4±2 days in patients with an occluded and non-occluded IRA before PCI. | At 4±2 days
Myocardial infarct size (as a percentage of myocardium at risk) both assessed by cardiac MRI at 4±2 days in the per protocol population who are cooled according to protocol and meet inclusion criteria. | At 4±2 days
Myocardial infarct size (as a percentage of myocardium at risk) both assessed by cardiac MRI at 4±2 days in patients with anterior or inferior myocardial infarctions separately. | At 4±2 days
The effect of the hypothermia protocol on the incidence of death. | 45±15 days and 6 months.
Plasma level of high sensitivity Troponin T AUC through 48 hours and peak plasma level of high sensitivity Troponin T within 48 hours after AMI. | 48 hours
ST-segment resolution 1.5 hour after opening the IRA. | 1.5 hours
Coronary blood flow and coronary angiography at the index event estimated by TIMI coronary flow and coronary perfusion grading. | 2 hours
Plasma NT-proBNP levels at day 4±2. | Day 4±2.
Incidence of death at 1, 2, 3, 4 and 5 years. | 5 years
Myocardial infarct size (as a percentage of myocardium at risk) assessed by cardiac MRI at 6±1 months. | 6 months
Incidence of heart failure within 45±15 days. | 6 months
Incidence of pulmonary oedema. | 1 week
Incidence of infections | 1 week
Incidence of bleedings | 1 week
The effect of the hypothermia protocol on the incidence of recurrent MI. | 6 months
The effect of the hypothermia protocol on the incidence of emergent stent revascularisation. | 6 months
The effect of the hypothermia protocol on the incidence of any hospitalisation. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Erlinge, MD PhD, Principal Investigator — Department of Cardiology, Skane University Hospital, Lund, Sweden; Göran K Olivecrona, MD PhD, Principal Investigator — Department of Cardiology, Skane University Hospital, Lund, Sweden; Anthony Mullins, Study Director — Philips Healthcare, San Diego, CA, USA; Lars Wallentin, MD PhD, Study Chair — Uppsala University Hospital, Uppsala, Sweden
Locations (10):
- Austria (3):
  - Graz University Hospital, Graz
  - Innsbruck University Hospital, Innsbruck
  - Medical University of Vienna, Vienna
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
- University Medical Centre, Ljubljana, Slovenia
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund, Sweden, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Nordlund D, Heiberg E, Carlsson M, Frund ET, Hoffmann P, Koul S, Atar D, Aletras AH, Erlinge D, Engblom H, Arheden H. Extent of Myocardium at Risk for Left Anterior Descending Artery, Right Coronary Artery, and Left Circumflex Artery Occlusion Depicted by Contrast-Enhanced Steady State Free Precession and T2-Weighted Short Tau Inversion Recovery Magnetic Resonance Imaging. Circ Cardiovasc Imaging. 2016 Jul;9(7):e004376. doi: 10.1161/CIRCIMAGING.115.004376. PMID 27412659
- [Derived] Engblom H, Tufvesson J, Jablonowski R, Carlsson M, Aletras AH, Hoffmann P, Jacquier A, Kober F, Metzler B, Erlinge D, Atar D, Arheden H, Heiberg E. A new automatic algorithm for quantification of myocardial infarction imaged by late gadolinium enhancement cardiovascular magnetic resonance: experimental validation and comparison to expert delineations in multi-center, multi-vendor patient data. J Cardiovasc Magn Reson. 2016 May 4;18(1):27. doi: 10.1186/s12968-016-0242-5. PMID 27145749
- [Derived] Tufvesson J, Carlsson M, Aletras AH, Engblom H, Deux JF, Koul S, Sorensson P, Pernow J, Atar D, Erlinge D, Arheden H, Heiberg E. Automatic segmentation of myocardium at risk from contrast enhanced SSFP CMR: validation against expert readers and SPECT. BMC Med Imaging. 2016 Mar 5;16:19. doi: 10.1186/s12880-016-0124-1. PMID 26946139
- [Derived] Erlinge D, Gotberg M, Noc M, Lang I, Holzer M, Clemmensen P, Jensen U, Metzler B, James S, Botker HE, Omerovic E, Koul S, Engblom H, Carlsson M, Arheden H, Ostlund O, Wallentin L, Klos B, Harnek J, Olivecrona GK. Therapeutic hypothermia for the treatment of acute myocardial infarction-combined analysis of the RAPID MI-ICE and the CHILL-MI trials. Ther Hypothermia Temp Manag. 2015 Jun;5(2):77-84. doi: 10.1089/ther.2015.0009. Epub 2015 May 18. PMID 25985169
- [Derived] Erlinge D, Gotberg M, Lang I, Holzer M, Noc M, Clemmensen P, Jensen U, Metzler B, James S, Botker HE, Omerovic E, Engblom H, Carlsson M, Arheden H, Ostlund O, Wallentin L, Harnek J, Olivecrona GK. Rapid endovascular catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. The CHILL-MI trial: a randomized controlled study of the use of central venous catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. J Am Coll Cardiol. 2014 May 13;63(18):1857-65. doi: 10.1016/j.jacc.2013.12.027. Epub 2014 Feb 5. PMID 24509284
- [Derived] Erlinge D, Gotberg M, Grines C, Dixon S, Baran K, Kandzari D, Olivecrona GK. A pooled analysis of the effect of endovascular cooling on infarct size in patients with ST-elevation myocardial infarction. EuroIntervention. 2013 Apr 22;8(12):1435-40. doi: 10.4244/EIJV8I12A217. PMID 23164721